CLINICAL TRIAL: NCT01117012
Title: An Open-Label, Rollover Study to Evaluate the Long Term Safety and Efficacy of VX-770 in Subjects With Cystic Fibrosis
Brief Title: Rollover Study of VX-770 in Cystic Fibrosis Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX08-770-105; PERSIST
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VX-770 (Experimental): VX-770 (ivacaftor) 150 milligram (mg) tablet orally twice daily (q12h).
  Interventions: Drug: Ivacaftor

INTERVENTIONS:
Drug: Ivacaftor
  Other Names: VX-770

SUMMARY:
The primary objective of the study was to evaluate the safety of long-term VX-770 treatment in participants with cystic fibrosis (CF). The secondary objective of the study was to evaluate the efficacy of long-term VX-770 treatment in subjects with CF.

DETAILED DESCRIPTION:
This open-label, rollover study of orally administered VX-770 was conducted in participants with CF to evaluate the safety and efficacy of long-term VX-770 treatment. Participants who were previously enrolled in Study 102 (VX08-770-102/NCT00909532) and Study 103 (VX08-770-103/NCT00909727), and met certain criteria were eligible to enroll in this study (Study 105/VX08-770-105/NCT01117012).

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have completed the assigned study treatment in Study 102 or Study 103
2. Participants who are females of childbearing potential must have a negative urine pregnancy test on Day 1 (first dose of VX-770)
3. Participants who are able to understand and comply with protocol requirements, restrictions, and instructions and likely to complete the study as planned, as judged by the investigator
4. Participants of child bearing potential and who are sexually active must meet the contraception requirements
5. Participants must sign the informed consent form (ICF), and where appropriate, assent must be obtained

Exclusion Criteria:

1. Participants with a history of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject
2. Participants with a history of study treatment intolerance as observed in their previous VX-770 study that, in the opinion of the investigator, might pose an additional risk in administering study drug to the subject
3. Participants who are pregnant, planning a pregnancy, breast-feeding, or not willing to follow contraception requirements
4. Participants taking any inhibitors or inducers of Cytochrome P450 3A4 (CYP3A4), including certain herbal medications (for example, St. John's Wort) and grapefruit/grapefruit juice

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward McKone, MD, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (58):
- United States (36):
  - Birmingham, Alabama
  - Oakland, California
  - Palo Alto, California
  - San Diego, California
  - Denver, Colorado
  - Atlanta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Long Branch, New Jersey
  - Buffalo, New York
  - New Hyde Park, New York
  - Syracuse, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Salt Lake City, Utah
  - Chrlottesville, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
- Australia (7):
  - Westmead, New South Wales
  - Chermside, Queensland
  - Herston, Queensland
  - South Brisbane, Queensland
  - Parkville, Victoria
  - Nedlands, Western Australia
  - Subiaco, Western Australia
- Canada (4):
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Montreal, Quebec
- Prague, Czechia
- France (2):
  - Paris
  - Roscoff
- Germany (4):
  - Erlangen
  - Jena
  - Munich
  - Würzburg
- Ireland (2):
  - Cork
  - Dublin
- United Kingdom (2):
  - Belfast, Northern Ireland
  - London

REFERENCES:
- [Derived] McKone EF, Borowitz D, Drevinek P, Griese M, Konstan MW, Wainwright C, Ratjen F, Sermet-Gaudelus I, Plant B, Munck A, Jiang Y, Gilmartin G, Davies JC; VX08-770-105 (PERSIST) Study Group. Long-term safety and efficacy of ivacaftor in patients with cystic fibrosis who have the Gly551Asp-CFTR mutation: a phase 3, open-label extension study (PERSIST). Lancet Respir Med. 2014 Nov;2(11):902-910. doi: 10.1016/S2213-2600(14)70218-8. Epub 2014 Oct 9. PMID 25311995

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Cystic Fibrosis (CF) who had completed the Study VX08-770-102 (Study 102/NCT00909532) and Study VX08-770-103 (Study 103/NCT00909727), were enrolled in this Study VX08-770-105 (Study 105/NCT01117012).
Pre-assignment Details: A total of 192 subjects were enrolled. Efficacy results are presented as per the treatment received in previous study (Placebo/Ivacaftor [VX-770]).
Groups:
- Placebo/VX-770: Participants who received placebo during the parent study (Study 102 or 103), received VX-770 150 milligram (mg) tablet orally twice daily (q12h).
- VX-770/VX-770: Participants who received VX-770 during the parent study (Study 102 or 103), received VX-770 150 mg tablet orally q12h.
Period: Overall Study
Arm/Group | Placebo/VX-770 | VX-770/VX-770
Started | 89 | 103
Completed | 81 | 98
Not Completed | 8 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Undefined | 4 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who were enrolled and received at least 1 dose of study drug during Study 105.
Groups:
- Placebo/VX-770: Participants who received placebo during the parent study (Study 102 or 103), received VX-770 150 mg tablet orally q12h.
- Total: Total of all reporting groups
Arm/Group | Placebo/VX-770 | VX-770/VX-770 | Total
Number analyzed (Participants) | 89 | 103 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.0 (10.94) | 23.2 (11.55) | 22.6 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 58 | 102
  Male | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-Serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse Event: any untoward medical occurrence in a participant during the study, including any unfavorable and unintended sign, symptom, or disease whether or not it was considered to be study drug related. This included any newly occurring event or previous condition that increased in severity or frequency after obtaining informed consent and assent (where applicable). SAE: medical event or condition, which resulted in any of following, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolonged hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect, important medical event. Non-Serious AEs included all AEs except SAEs.
Time Frame: Study 105: Day 1 up to Week 168
Population: Safety Set included all participants who received at least 1 dose of study drug during Study 105.
Measure: Number; unit: participants
Groups:
- VX-770: All participants who received VX-770 150 mg tablet orally q12h in Study 105.
Arm/Group | VX-770
Number analyzed (Participants) | 192
participants
  Non-Serious AEs | 190
  SAEs | 70

2. Secondary Outcome: Annualized Rate of Decline From Study 105 Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through Week 96
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Predicted FEV1 (for age, gender, and height) was calculated using the Knudson method. Baseline was defined as Study 105 Day 15.
Time Frame: Study 105: Baseline through Week 96
Population: Full Analysis Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted of FEV1 per year
Arm/Group | Placebo/VX-770 | VX-770/VX-770
Number analyzed (Participants) | 89 | 103
percent predicted of FEV1 per year | -0.30 [-2.47 to 1.86] | -1.23 [-2.10 to -0.35]

3. Secondary Outcome: Absolute Change From Study 105 Baseline in Percent Predicted FEV1 Through Week 96
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Predicted FEV1 (for age, gender, and height) was calculated using the Knudson method. Baseline was defined as the most recent measurement prior to intake of the first dose of study drug in Study 105. Absolute Change at Week 48 and Week 96 are reported.
Time Frame: Study 105: Baseline through Week 96
Population: Full Analysis Set. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure and n signifies participants who were evaluable for specified categories for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percent predicted of FEV1
Arm/Group | Placebo/VX-770 | VX-770/VX-770
Number analyzed (Participants) | 85 | 99
percent predicted of FEV1
  Absolute Change at Week 48 (n = 85, 99) | 9.2585 (9.63822) | -0.4422 (8.62332)
  Absolute Change at Week 96 (n = 76, 97) | 9.8194 (11.22812) | 0.1581 (9.01629)

4. Secondary Outcome: Absolute Change From Study 105 Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score Through Week 96
Description: The CFQ-R is a validated patient-reported outcome measuring health-related quality of life for subjects with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Absolute Change at Week 48 and Week 96 are reported.
Time Frame: Study 105: Baseline through Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/VX-770 | VX-770/VX-770
Number analyzed (Participants) | 86 | 99
units on a scale
  Absolute Change at Week 48 (n = 86, 99) | 7.43 (16.600) | -1.94 (16.550)
  Absolute Change at Week 96 (n = 77, 97) | 10.05 (15.254) | 0.77 (14.305)

5. Secondary Outcome: Annualized Pulmonary Exacerbation Event Rate
Description: Annualized event rate was calculated by regression with negative binomial distribution.
Time Frame: Study 105: Day 1 through Week 96
Population: Full Analysis Set.
Measure: Number; unit: events per year
Arm/Group | Placebo/VX-770 | VX-770/VX-770
Number analyzed (Participants) | 89 | 103
events per year | 0.463 | 0.658

6. Secondary Outcome: Annualized Duration of Pulmonary Exacerbation Events
Time Frame: Study 105: Day 1 through Week 96
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: Days per year
Arm/Group | Placebo/VX-770 | VX-770/VX-770
Number analyzed (Participants) | 89 | 103
Days per year | 10.89 (20.124) | 17.27 (30.974)

7. Secondary Outcome: Absolute Change From Study 105 Baseline in Weight Through Week 96
Description: Weight is a measurement of nutritional status. Absolute change in weight, measured in kilograms (kg), at Week 48 and Week 96 are reported.
Time Frame: Study 105: Baseline through Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo/VX-770 | VX-770/VX-770
Number analyzed (Participants) | 86 | 99
kg
  Absolute Change at Week 48 (n = 86, 99) | 4.03 (3.677) | 1.26 (3.844)
  Absolute Change at Week 96 (n = 76, 97) | 4.93 (5.577) | 2.62 (5.909)

ADVERSE EVENTS:
Time Frame: Study 105: Day 1 through Week 168
Arm/Group | VX-770
Serious Adverse Events (participants affected / at risk) | 70/192
Other Adverse Events (participants affected / at risk) | 190/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VX-770 (N=192)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 42
Influenza (Infections and infestations) | 4
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Aspergilloma (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Lung infection pseudomonal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 1
Distal ileal obstruction syndrome (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Chest X-ray abnormal (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Pulmonary function test decreased (Investigations) | 1
Headache (Nervous system disorders) | 2
Hemiplegic migraine (Nervous system disorders) | 1
Hypoglycaemic seizure (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Affective disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Depression suicidal (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Vestibular disorder (Ear and labyrinth disorders) | 1
Device occlusion (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Renal tubular disorder (Renal and urinary disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VX-770 (N=192)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 94
Upper respiratory tract infection (Infections and infestations) | 65
Nasopharyngitis (Infections and infestations) | 39
Sinusitis (Infections and infestations) | 29
Gastroenteritis (Infections and infestations) | 13
Rhinitis (Infections and infestations) | 10
Influenza (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 9
Respiratory tract infection viral (Infections and infestations) | 8
Tonsillitis (Infections and infestations) | 8
Oral candidiasis (Infections and infestations) | 7
Respiratory tract infection (Infections and infestations) | 7
Bronchitis (Infections and infestations) | 6
Candidiasis (Infections and infestations) | 6
Gastroenteritis viral (Infections and infestations) | 6
Viral upper respiratory tract infection (Infections and infestations) | 6
Oral herpes (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 5
Vulvovaginal mycotic infection (Infections and infestations) | 5
Bacterial disease carrier (Infections and infestations) | 4
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 4
Ear infection (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Acute sinusitis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 3
Cystitis (Infections and infestations) | 3
Otitis media (Infections and infestations) | 3
Pseudomonas infection (Infections and infestations) | 3
Tooth abscess (Infections and infestations) | 3
Viral infection (Infections and infestations) | 3
Conjunctivitis infective (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Oropharyngeal candidiasis (Infections and infestations) | 2
Otitis externa (Infections and infestations) | 2
Tracheobronchitis (Infections and infestations) | 2
Vulvovaginal candidiasis (Infections and infestations) | 2
Alveolar osteitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Body tinea (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Erythema migrans (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastritis viral (Infections and infestations) | 1
Genital candidiasis (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Genital infection fungal (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes simplex ophthalmic (Infections and infestations) | 1
Infection parasitic (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Lower respiratory tract infection viral (Infections and infestations) | 1
Mycobacterial infection (Infections and infestations) | 1
Nail bed infection bacterial (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Rhinotracheitis (Infections and infestations) | 1
Serratia infection (Infections and infestations) | 1
Vaginitis bacterial (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 86
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 39
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 26
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 24
Productive cough (Respiratory, thoracic and mediastinal disorders) | 24
Rales (Respiratory, thoracic and mediastinal disorders) | 19
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 17
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 14
Wheezing (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 9
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 9
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 8
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 5
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 4
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 4
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 3
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 2
Nasal turbinate abnormality (Respiratory, thoracic and mediastinal disorders) | 2
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 23
Constipation (Gastrointestinal disorders) | 22
Diarrhoea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 21
Abdominal pain upper (Gastrointestinal disorders) | 19
Nausea (Gastrointestinal disorders) | 19
Dyspepsia (Gastrointestinal disorders) | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9
Flatulence (Gastrointestinal disorders) | 6
Toothache (Gastrointestinal disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 5
Rectal haemorrhage (Gastrointestinal disorders) | 4
Distal ileal obstruction syndrome (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Steatorrhoea (Gastrointestinal disorders) | 2
Duodenitis (Gastrointestinal disorders) | 1
Gastric hypomotility (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Tooth impacted (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Bacterial test positive (Investigations) | 16
Weight decreased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 9
Pulmonary function test decreased (Investigations) | 8
Alanine aminotransferase increased (Investigations) | 6
Fungal test positive (Investigations) | 6
Glucose urine present (Investigations) | 6
Vitamin D decreased (Investigations) | 6
Blood glucose increased (Investigations) | 5
Prothrombin time prolonged (Investigations) | 5
Gamma-glutamyltransferase increased (Investigations) | 4
Hepatic enzyme increased (Investigations) | 4
Liver function test abnormal (Investigations) | 4
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 3
Culture throat positive (Investigations) | 3
Forced expiratory volume decreased (Investigations) | 3
White blood cell count increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood glucose decreased (Investigations) | 2
Blood iron decreased (Investigations) | 2
Blood urine present (Investigations) | 2
Body temperature increased (Investigations) | 2
Breath sounds abnormal (Investigations) | 2
Cardiac murmur (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 2
Eosinophil count increased (Investigations) | 2
Neutrophil count increased (Investigations) | 2
Platelet count increased (Investigations) | 2
Protein urine present (Investigations) | 2
Spirometry abnormal (Investigations) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Blood albumin increased (Investigations) | 1
Blood bilirubin unconjugated increased (Investigations) | 1
Blood calcium increased (Investigations) | 1
Blood cortisol increased (Investigations) | 1
Blood immunoglobulin E increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Clostridium test positive (Investigations) | 1
Coagulation factor increased (Investigations) | 1
Electrocardiogram T wave peaked (Investigations) | 1
Gastrointestinal examination abnormal (Investigations) | 1
Glycosylated haemoglobin increased (Investigations) | 1
Haemoglobin increased (Investigations) | 1
Monocyte count increased (Investigations) | 1
Nitrite urine present (Investigations) | 1
Peak expiratory flow rate decreased (Investigations) | 1
Serum ferritin decreased (Investigations) | 1
Sputum abnormal (Investigations) | 1
Urine leukocyte esterase (Investigations) | 1
Urine leukocyte esterase positive (Investigations) | 1
Weight increased (Investigations) | 1
Headache (Nervous system disorders) | 45
Dizziness (Nervous system disorders) | 12
Sinus headache (Nervous system disorders) | 7
Hypoaesthesia (Nervous system disorders) | 5
Lethargy (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 4
Migraine (Nervous system disorders) | 3
Convulsion (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Ageusia (Nervous system disorders) | 1
Burning sensation (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Pyrexia (General disorders) | 35
Fatigue (General disorders) | 13
Catheter site pain (General disorders) | 7
Chest pain (General disorders) | 6
Influenza like illness (General disorders) | 6
Non-cardiac chest pain (General disorders) | 6
Pain (General disorders) | 5
Chills (General disorders) | 3
Malaise (General disorders) | 3
Oedema peripheral (General disorders) | 3
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 2
Injection site pain (General disorders) | 2
Adverse drug reaction (General disorders) | 1
Catheter site swelling (General disorders) | 1
Drug interaction (General disorders) | 1
Exercise tolerance decreased (General disorders) | 1
Infusion site pain (General disorders) | 1
Medical device pain (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 26
Back pain (Musculoskeletal and connective tissue disorders) | 14
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Clubbing (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 13
Acne (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4
Night sweats (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3
Sunburn (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 2
Rash papular (Skin and subcutaneous tissue disorders) | 2
Skin wrinkling (Skin and subcutaneous tissue disorders) | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 5
Laceration (Injury, poisoning and procedural complications) | 4
Ligament sprain (Injury, poisoning and procedural complications) | 4
Contusion (Injury, poisoning and procedural complications) | 3
Arthropod sting (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 2
Hand fracture (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 2
Meniscus lesion (Injury, poisoning and procedural complications) | 2
Muscle strain (Injury, poisoning and procedural complications) | 2
Skeletal injury (Injury, poisoning and procedural complications) | 2
Wrist fracture (Injury, poisoning and procedural complications) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Muscle injury (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1
Stab wound (Injury, poisoning and procedural complications) | 1
Sternal injury (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Tongue injury (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 5
Glucose tolerance impaired (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Iron deficiency (Metabolism and nutrition disorders) | 2
Vitamin K deficiency (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypovitaminosis (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Insulin resistance (Metabolism and nutrition disorders) | 1
Lactose intolerance (Metabolism and nutrition disorders) | 1
Vitamin A deficiency (Metabolism and nutrition disorders) | 1
Zinc deficiency (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 11
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Sleep disorder (Psychiatric disorders) | 2
Abnormal dreams (Psychiatric disorders) | 1
Adjustment disorder (Psychiatric disorders) | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1
Mood swings (Psychiatric disorders) | 1
Phagophobia (Psychiatric disorders) | 1
Ear pain (Ear and labyrinth disorders) | 6
Vertigo (Ear and labyrinth disorders) | 4
Cerumen impaction (Ear and labyrinth disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Ear pruritus (Ear and labyrinth disorders) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1
Conjunctivitis (Eye disorders) | 5
Vision blurred (Eye disorders) | 3
Conjunctivitis allergic (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Lens disorder (Eye disorders) | 1
Meibomian gland dysfunction (Eye disorders) | 1
Myopia (Eye disorders) | 1
Ocular vascular disorder (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Seasonal allergy (Immune system disorders) | 9
Drug hypersensitivity (Immune system disorders) | 3
Hypersensitivity (Immune system disorders) | 3
Allergy to animal (Immune system disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 6
Breast mass (Reproductive system and breast disorders) | 1
Cervix inflammation (Reproductive system and breast disorders) | 1
Dyspareunia (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Haematuria (Renal and urinary disorders) | 4
Nephrolithiasis (Renal and urinary disorders) | 3
Polyuria (Renal and urinary disorders) | 2
Cystitis interstitial (Renal and urinary disorders) | 1
Glycosuria (Renal and urinary disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 5
Coagulopathy (Blood and lymphatic system disorders) | 1
Neutrophilia (Blood and lymphatic system disorders) | 1
Polycythaemia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 1
Intracardiac thrombus (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 3
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 4
Cataract congenital (Congenital, familial and genetic disorders) | 1
Cystic fibrosis pancreatic (Congenital, familial and genetic disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Adrenal suppression (Endocrine disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days